CLINICAL TRIAL: NCT03140956
Title: Pharmacokinetics of Levodopa After Repeated Doses of Different Pellet Formulations; An Open, Randomized Study With Crossover Design in Healthy Male Subjects
Brief Title: Pharmacokinetic of Levodopa Study in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3112006
Record Dates: First submitted 2017-04-12; First posted 2017-05-04 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Levodopa formulation D (Experimental): Levodopa formulation D
  Interventions: Drug: Levodopa, carbidopa, ODM-104
- Levodopa formulation E (Experimental): Levodopa formulation E
  Interventions: Drug: Levodopa, carbidopa, ODM-104
- Levodopa formulation F (Experimental): Levodopa formulation F
  Interventions: Drug: Levodopa, carbidopa, ODM-104
- Sinemet IR 100/25mg (Active Comparator): Sinemet IR 100/25MG
  Interventions: Drug: Levodopa, carbidopa, ODM-104
- Sinemet CR 100/25mg (Active Comparator): Sinemet IR 100/25MG
  Interventions: Drug: Levodopa, carbidopa, ODM-104
- ODM-104 100mg (Experimental): ODM-104 100MG
  Interventions: Drug: Levodopa, carbidopa, ODM-104
- Carbidopa 20mg (Active Comparator): Carbidopa 20MG
  Interventions: Drug: Levodopa, carbidopa, ODM-104
- Carbidopa 65mg (Active Comparator): Carbidopa 65MG
  Interventions: Drug: Levodopa, carbidopa, ODM-104

INTERVENTIONS:
Drug: Levodopa, carbidopa, ODM-104 — Crossover design. Study treatments will be administered in randomized order 4 times a day.
  Other Names: Sinemet

SUMMARY:
The purpose of the study is to investigate PK of levodopa in plasma after repeated doses of 3 levodopa formulations given in combination with carbidopa and ODM-104 and compared to the PK of standard IR and CR levodopa formulations in the same combination.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Finnish speaking males between 18-65 years of age.
* Body mass index (BMI) between 19-32 kg/m2 (BMI = weight/height2).
* Weight at least 60 kg.
* Regular intestinal transit (no recent history of recurrent constipation, diarrhoea, or other intestinal problems, and no history of major gastrointestinal surgery).
* Sexually active study subjects, unless surgically sterile must adhere to a proper form of contraception (hormonal contraception or intrauterine device on female partner and an additional barrier method used at least by one of the partners) and must not donate sperm from the first study treatment administration until 3 months after the last study treatment administration.

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic, endocrine, neurological or psychiatric disease or cancer (except local non-melanoma skin cancer) within the previous 2 years.
* Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study. As an exception, paracetamol for occasional pain is allowed.
* Any clinically significant abnormal laboratory value or ECG (such as prolonged QTcF > 450 ms or QRS > 120 ms) that in the opinion of the investigator could interfere with the interpretation of study results or cause a health risk for the subject if he takes part in the study.
* Known hypersensitivity to the active substances or the excipients of the drugs.
* History of vasovagal collapses or vagal reactions with unexplained reason within the previous 2 years or a tendency for vasovagal reactions during blood sampling.
* HR < 40 beats per minute (bpm) or > 90 bpm in the supine position after 5 min rest at the screening visit.
* At the screening visit:systolic BP < 90 mmHg or > 150 mmHg in the supine position after 5 min rest and diastolic BP < 50 mmHg or > 90 mmHg in the supine position after 5 min rest.
* History of anaphylactic/anaphylactoid reactions.
* Strong tendency to motion sickness.
* Recent or current (suspected) drug abuse.
* Recent or current alcohol abuse; regular drinking of more than 21 units per week (1 unit = 4 cl spirits or equivalent).
* Current use of nicotine containing products more than 5 cigarettes (or equivalent)/day and/or inability to refrain from the use of nicotine containing products during the study (from the screening visit to the end-of-study visit).
* Use of caffeine containing beverages more than 600 mg of caffeine/day and/or inability to refrain from using caffeine containing beverages 10 h before and during the study periods.
* Blood donation or loss of a significant amount of blood within 90 days before the first study treatment administration.
* Participation in an investigational drug study or administration of an investigational drug within 90 days before the first study treatment administration.
* Unsuitable veins for repeated venipuncture or cannulation.
* Predictable poor compliance or inability to communicate well with the study centre personnel.
* Inability to participate in all treatment periods.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax) of levodopa | 24 hours
  Peak Plasma Concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology Unit, Orion Pharma, Espoo, Finland